CLINICAL TRIAL: NCT03393962
Title: Interventional Treatment of Ovarian Cancer With Cancer Antigen-specific Engineered Immune Effector T Lymphocytes (OC-EIEs)
Brief Title: Intervention of Ovarian Cancer With Antigen-specific Engineered Immune Effectors
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: combine with another trial
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17024
Record Dates: First submitted 2017-12-28; First posted 2018-01-09 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Cytotoxic lymphocyte; Cancer specific antigen
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OC-EIEs (Experimental): Autologous ovarian cancer antigen-specific cytotoxic lymphocytes
  Interventions: Biological: OC-EIEs

INTERVENTIONS:
Biological: OC-EIEs — 2 to 4 infusions, once a week, 0.1~4x10^6 CTLs/kg; injection via IV, abdominal cavity or intrastumoral.

SUMMARY:
This is a single-arm, open-label, phase I/II trial to evaluate the safety and efficacy of ovarian cancer-specific, engineered immune effectors (OC-EIEs) in women.

DETAILED DESCRIPTION:
Ovarian cancer (OC) is a cancer that is derived from an ovary. The majority of OC arises from the epithelium (outer lining) of the ovary. In 2015, OC was found in 1.2 million women and resulted in 161,100 deaths worldwide. Among women, OC is the seventh-most common cancer and the eighth-most common cause of cancer death. Treatment for OC consists of surgery, chemotherapy, immunotherapy and radiotherapy. The kind of treatment depends on many factors, including the type of OC, its stage and grade, as well as the general health of the patient.

Adoptive immunotherapy with cytotoxic T lymphocytes (CTLs) reactive with tumor antigens has proven to be effective against many types of cancer. OC has been shown to be highly immunogenic and therefore may respond well to innovative antigen-specific immunotherapy. Here, through cancer antigen screening and careful target antigen evaluation, the investigation aims to evaluate the safety and efficacy of multiple infusions of OC antigen-specific, engineered immune effectors (EIEs) in patients with OC.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent obtained prior to any study-specific procedures.
2. Age older than 10 years.
3. Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
4. Expected survival ≥ 12 weeks.
5. Histologically confirmed and documented high risk International Federation of Gynecology and Obstetrics (FIGO): Stage II-IV.
6. Not pregnant, and on appropriate birth control of childbearing potential.
7. Initial hematopoietic reconstitution with

   * neutrophils (ANC) ≥ 1,000/mm^3;
   * platelet (PLT) ≥ 100,000/mm^3.
8. Proper renal and hepatic functions (ULN denotes "upper limit of normal range") with

   * serum creatinine ≤ 2×ULN;
   * serum bilirubin ≤ 2×ULN;
   * AST/ALT ≤ 2×ULN;
   * ALKP ≤ 5×ULN;
   * serum bilirubin. 2.0 is acceptable in the setting of known Gilbert's syndrome.
9. Human immunodeficiency virus (HIV) and hepatitis C virus (HCV) test negative.

Exclusion Criteria:

1. Patients with ovarian tumors with low malignant potential (i.e. borderline tumors);
2. Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure (prior, current or planned treatment).
3. Prior treatment of any adoptive T cell therapy.
4. Current or recent treatment (within the 14-day period prior to Day 0) with any immune suppressive drug
5. Minor surgical procedures within 2 days prior to Day 0 (including central venous access device placement for chemotherapy administration, tumor biopsies, needle aspirations).
6. Pregnant or lactating females.
7. Inadequate bone marrow function with

   * absolute neutrophil count < 1,000/mm^3;
   * platelet count < 100,000/mm^3;
   * Hb < 9 g/dL.
8. Inadequate liver and renal function with

   * serum (total) bilirubin > 1.5 x ULN;
   * AST & ALT > 2.5 x ULN (> 5 x ULN in patients with liver metastases);
   * alkaline phosphatase > 2.5 x ULN;
   * serum creatinine >2.0 mg/dl (> 177 μmol/L);
   * urine dipstick for protein uria should be < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < 1 g of protein/24 hr.
9. Serious active infection requiring i.v. antibiotics
10. Subject infected with HCV (HCV antibody positive), or HIV (HIV antibody positive),Treponema pallidum antibody positive or TB culture positive.

Ages: 10 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety of OC-EIEs in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 6 months
  percentage of patients with grade 3 or above adverse effect

SECONDARY OUTCOMES:
Expansion of OC-EIEs | 8 weeks.
  The increased fold of specificity of OC-EIEs, will be analyzed by enzyme-linked immunospot assay (ELISPOT)
percentage of complete response | 1 year
  Objective response will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
percentage of partial response | 1 year
  Objective response will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
percentage of stable disease | 1 year
  Objective response will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
percentage of progressive disease | 1 year
  Objective response will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute; Qichun Cai, MD, Study Director — Jinshazhou Hospital of Guangzhou University of Chinese Medicine; Xun Lai, MD, Study Director — Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center
Locations (3):
- China (3):
  - Jinshazhou Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No